CLINICAL TRIAL: NCT04666688
Title: A Phase 1/2 Open-label, Multi-center Study of the Safety, Pharmacokinetics, and Anti-tumor Activity of LYT-200 as a Single Agent and in Combination With Chemotherapy or Tislelizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: LYT-200 Alone and in Combination With Chemotherapy or Tislelizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PureTech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LYT-200-2020-01
Record Dates: First submitted 2020-11-25; First posted 2020-12-14 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Cancer; Solid Tumor; Pancreatic Cancer; Urothelial Carcinoma; Head and Neck Cancer; Colorectal Cancer
Keywords: Metastatic cancer; Solid tumors; Combination therapy; Pancreatic cancer; Colon cancer; Bile duct cancer; Urothelial Carcinoma; Head and Neck Cancer; Colorectal Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Pancreatic Neoplasms; Carcinoma, Transitional Cell; Head and Neck Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Bile Duct Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: Phase 1/2, two part, open-label study, which will enroll Part 1 and Part 2 sequentially. Part 1 is a single agent dose escalation design utilizing a continuous reassessment method (CRM) and a combination portion using a 4+2 study design. Part 2 is dose expansion into specific disease indications based on outcomes from Part 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 single agent dose escalation (Experimental): LYT-200 in metastatic solid tumors
  Interventions: Drug: LYT-200
- Part 1 combination agents dose expansion (Experimental): LYT-200 in combination with chemotherapy or Tislelizumab in select metastatic solid tumors
  Interventions: Drug: LYT-200; Drug: Tislelizumab; Drug: Gemcitabine/nab-paclitaxel
- Part 2 (Experimental): LYT-200 combination dose expansion in select metastatic solid tumors based on outcomes of Part 1
  Interventions: Drug: LYT-200; Drug: Tislelizumab; Drug: Gemcitabine/nab-paclitaxel

INTERVENTIONS:
Drug: LYT-200 — monoclonal antibody (mAb), targeting galectin-9 protein
Drug: Tislelizumab — anti-PD-1 monoclonal antibody
  Arms: Part 1 combination agents dose expansion; Part 2
Drug: Gemcitabine/nab-paclitaxel — chemotherapy
  Arms: Part 1 combination agents dose expansion; Part 2

SUMMARY:
A Phase 1/2 Open-label, Multi-center Study of the Safety, Pharmacokinetics, and Anti-tumor Activity of LYT-200 Alone and in Combination with Chemotherapy or Tislelizumab in Patients with Metastatic Solid Tumors

DETAILED DESCRIPTION:
This is an open-label, uncontrolled, multicenter Phase 1/2 study with a dose escalation phase (Part 1) and a cohort expansion phase (Part 2) in patients with relapsed/refractory metastatic solid tumors.

Part 1: Dose Escalation Phase_Single Agent A dose-finding study will be conducted using a continuous reassessment method (CRM) to establish dose-limiting toxicities (DLTs) and the recommended Phase 2 dose (RP2D).

Part 1: Dose Escalation Phase_Combination A dose-finding combination study with chemotherapy or tislelizumab will be conducted using a 4+2 study design to establish dose-limiting toxicities (DLTs) and the recommended Phase 2 dose (RP2D).

Part 2: The second part of the protocol will be a dose expansion in both/or either single agent or combination based on the RP2D determined in Part 1, in patients with metastatic/advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Part 1

1. Written Informed Consent (mentally competent patient, able to understand and willing to sign the informed consent form)
2. Age ≥ 18 years, male or non-pregnant female
3. Able to comply with the study protocol, as per Investigator's judgment
4. Histologically confirmed, unresectable locally advanced or metastatic cancer. There are no limits to prior lines of therapies received for the treatment of the cancer condition for which the patient is being enrolled into this study.

   1. For the Part 1 combination urothelial carcinoma Cohorts 13 and 14: histologically or cytologically confirmed diagnosis of unresectable, locally advanced or metastatic urothelial carcinoma of the renal pelvis, ureter, bladder, or urethra (i.e., transitional cell carcinoma).
   2. For the Part 1 combination H/N cancer Cohorts 11 and 12: histologically confirmed, locally advanced or metastatic squamous cell carcinoma of head and neck (SCCHN; oral cavity, oropharynx, hypopharynx, or larynx).
5. For urothelial and H/N combination cancer cohorts, prior exposure to immunotherapy is allowed, with standard of care treatment options and/or within a clinical trial context. If the patient received an anti-PD-1 and/or an anti-PD-L1 containing regimen at any point, they must have demonstrated at least stable disease, as per RECIST 1.1 or iRECIST criteria to one of these treatment regimens, if these measurements are available. If RECIST or iRECIST measurements are not available, then clinical PFS of at least 4 months is required to have been achieved on any of the prior anti-PD-1 and/or anti-PD-L1 containing regimens.
6. There is no PD-L1 expression requirement for the Part 1 combination urothelial and H/N cohorts; however, fresh biopsy or archival tissue is required for assessment of PD-L1 by IHC, or a historical PD-L1 expression by IHC must be available. If PD-L1 expression data are already available, this does not override the protocol preference for obtaining a fresh biopsy whenever feasible.
7. For Part 1 combination cohort H/N cancer patients of oropharynx origin: human papilloma virus (HPV) status needs to be established in the screening period or at any point while patient is on study drug, unless it is historically known. p16+ as a surrogate for HPV+, HPV RNA ISH or DNA PCR are all acceptable. The study accepts both HPV+ and HPV- patients.
8. Life expectancy > 3 months according to Investigator's judgment
9. ECOG performance status 0-1
10. Patient able and willing to undergo pre- and on/post treatment biopsies. According to the Investigator's judgment, the planned biopsies should not expose the patient to substantially increased risk of complications. Every effort will be made that the same lesion is biopsied on repeat biopsies. If the patient is eligible according to all other criteria but declines to consent to a biopsy or there are other medical reasons precluding biopsy, this will be discussed with the Sponsor.
11. Measurable disease, according to RECIST v1.1. Note that lesions intended to be biopsied should not be target lesions.
12. Adequate hematologic and end organ function, defined by the following laboratory results obtained prior to first dose of study drug treatment, provided no anticancer treatment was administered within the last 7 days:

    1. neutrophil count ≥ 1 x 109/L
    2. platelet count ≥ 100 x 109/L; for hepatocellular carcinoma (HCC) in Part 1 ≥ 50 x 109/L
    3. hemoglobin ≥ 9.0 g/dL without transfusion in the previous week
    4. creatinine ≤ 1.5 x the upper limit of normal (ULN); or eGFR > 50 mg/mmol
    5. aspartate aminotransferase AST (SGOT) ≤ 3 x ULN (≤ 5 x ULN when HCC or hepatic metastases are present)
    6. alanine aminotransferase (ALT [SGPT]) ≤ 3 x ULN (≤ 5 x ULN when HCC or hepatic metastases present)
    7. bilirubin ≤ 1.5 x ULN (patients with known Gilbert's disease may have a bilirubin ≤ 3.0 x ULN)
    8. albumin ≥ 3.0 g/dL
    9. international normalized ratio (INR) and partial thromboplastin time (PTT) ≤ 1.5 x ULN, unless patient receiving anticoagulant therapy
13. No evidence of active serious infection or infections requiring parenteral antibiotics.
14. Women of childbearing potential must have a negative pregnancy test within 72 h prior to start of treatment. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or to use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 180 days after the last study treatment.

    A woman is of childbearing potential if she is post-menarche, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

    Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptom-thermal, or post ovulation methods) and withdrawal are not acceptable methods of contraception. Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists.
15. Four (4) weeks or 5 half-lives (whichever is shorter) since the last dose of anticancer therapy before the first LYT-200 administration
16. Bisphosphonate treatment (e.g., zoledronic acid) or denosumab are allowed if previously used prior to commencement of clinical trial.
17. Patients:

    1. who have already received at least one prior line of systemic therapy for metastatic or locally advanced disease, and/or
    2. who have a tumor type for which there are no available standard of care options
18. Patients who have not previously received a gemcitabine-containing regimen

Exclusion Criteria

1. Patient unwilling or unable to follow protocol requirements
2. Patient diagnosed with metastatic cancer of an unknown primary
3. Current illicit drug addiction (medical and recreational marijuana/cannabidiol [CBD]/ tetrahydrocannabinol [THC] would not be considered "illicit")
4. Clinically significant, active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease). Prophylactic or therapeutic use of anticoagulants is allowed.
5. Pregnant and/or lactating females
6. Receiving any other investigational agents or participating in any other clinical trial involving another investigational agent for treatment of solid tumors within 3 weeks or 5 half-lives of the administered drug (whichever is shorter) prior to the first dose of study drug, or major surgery or planned surgery within 4 weeks of the first dose of study drug (this includes dental surgery).
7. Radiation therapy within 4 weeks of the first dose of study drug, except for palliative radiotherapy to a limited field, such as for the treatment of bone pain or a focally painful tumor mass, and which does not jeopardize required measurable lesions for response assessment (RECIST v1.1).
8. Patients with fungating tumor masses
9. History or current evidence of any condition, therapy, any active infections, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator
10. Grade 4 immune-mediated toxicities with a prior checkpoint inhibitor. Grade 2 or Grade 3 pneumonitis or any other Grade 3 checkpoint inhibitor-related toxicity that led to immunotherapy treatment discontinuation. Low-grade (< Grade 3) toxicities, such as neuropathy from prior treatments, manageable electrolyte abnormalities and lymphopenia, alopecia and vitiligo are allowed.
11. History of other prior or other concomitant malignancy that requires other active treatment.
12. Active parenchymal brain metastases, patients with carcinomatous meningitis or leptomeningeal metastases. Patients with brain metastases are eligible provided they have shown clinically and radiographically stable disease for at least 4 weeks after definitive therapy and have not used steroids (> 10 mg/day of prednisone or equivalent) for at least 4 weeks prior to the first dose of study drug
13. Evidence of severe or uncontrolled systemic diseases, congestive heart failure > New York Heart Association (NYHA) class 2, myocardial infarction (MI) within 6 months, or laboratory finding that in the view of the Investigator makes it undesirable for the patient to participate in the trial
14. Any medical condition that the Investigator considers significant to compromise the safety of the patient or that impairs the interpretation of LYT-200 toxicity assessment
15. Serious non-healing wound, active ulcer, or untreated bone fracture unless for e.g., a rib fracture for (which does not elicit treatment)
16. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures. For the purposes of this study, "recurrent" is defined as ³ 3 drains in the last 30 days
17. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
18. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of Cycle 1, Day 1
19. History of pulmonary embolism, stroke or transient ischemic attack within 3 months prior to Cycle 1, Day 1
20. Active autoimmune disorder (except type I/II diabetes, hypothyroidism requiring only hormone replacement, vitiligo, psoriasis, or alopecia areata).
21. Requires systemic immunosuppressive treatment, including, but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (anti-TNF) agents. Patients who have received or are receiving acute, low dose systemic immunosuppressant medications (e.g., ≤ 10 mg/day of prednisone or equivalent) may be enrolled. Replacement therapy (e.g., thyroxine, insulin, physiologic corticosteroid replacement therapy [e.g., ≤ 10 mg/day of prednisone equivalent] for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone), topical steroids, intranasal steroids, intra-articular, and ophthalmic steroids is allowed.
22. Severe tumor-related pain (Grade 3, CTCAE v.5.0) unresponsive to broad analgesic interventions (oral and/or patches)
23. Hypercalcemia (defined as ³ Grade 3, per CTCAE v 5.0) despite use of bisphosphonates
24. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk of treatment complications
25. Received organ transplant(s)
26. Patients undergoing dialysis
27. For Part 1, hormonal androgen deprivation therapy is allowed to continue for patients with metastatic castration-resistant prostate cancer
28. Any ablative therapy (Radio Frequency Ablation or Percutaneous Ethanol Injection) for HCC < 6 weeks prior trial entry
29. Hepatic encephalopathy or severe liver adenoma
30. Child-Pugh score ≥ 7

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence of Treatment-Emergent Adverse Events [Safety] | approximately 1 year
  Evaluation of safety parameters including treatment emergent adverse events as detected by hematology, chemistry, coagulation safety labs, physical exams, vital signs, ECG, ECHO/MUGA, ECOG status.
Part 1: Incidence of Dose Limiting Toxicities [Tolerability] | approximately 1 year
  Evaluation of tolerability parameters including dose limiting toxicities as detected by hematology, chemistry, coagulation safety labs, physical exams, vital signs, ECG, ECHO/MUGA, ECOG status
Part 2: PFS or ORR [Preliminary Efficacy] | approximately 1 year
  PFS or ORR depending on tumor type

SECONDARY OUTCOMES:
Part 1: Pharmacokinetic (PK) profile of LYT-200: Maximum Plasma Concentration [Cmax] | approximately 1 year
  To characterize Cmax of LYT- 200
Part 1: Pharmacokinetic (PK) profile of LYT-200: Time to Maximum Plasma Concentraton [Tmax] | approximately 1 year
  To characterize Tmax of LYT- 200
Part 1: Pharmacokinetic (PK) profile of LYT-200: Area Under the Curve [AUC] | approximately 1 year
  To characterize AUC of LYT- 200
Part 1: Pharmacodynamics (PD) of LYT- 200 | approximately 1 year
  blood and tumor tissue sampling, cell and non-cell based, immunological and cancer related PD markers

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Filipovic, MD, Ph.D., Study Director — PureTech Health
Locations (12):
- United States (12):
  - UCLA, Los Angeles, California
  - University of Colorado Hospital, Denver, Colorado
  - Sarah Cannon Research Institute at Health One, Denver, Colorado
  - Sarah Cannon Research Institute, Florida Cancer Specialists, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics, Grand Rapids, Michigan
  - Columbia University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Tennessee Oncology, Nashville, Tennessee
  - University of Texas, M.D. Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas